CLINICAL TRIAL: NCT03006250
Title: The Effect of Desflurane vs Sevoflurane on Perioperative Respiratory Complications in Laryngeal Mask Airway Anesthesia: A Prospective Randomized Double-blinded Control Study
Brief Title: The Effect of Desflurane vs Sevoflurane on Perioperative Respiratory Complications in Laryngeal Mask Airway Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 15072016
Record Dates: First submitted 2016-07-24; First posted 2016-12-30 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia; Adverse Effect; Laryngeal Masks; Respiratory System Abnormalities
Keywords: Desflurane; Sevoflurane; Respiratory Complications
MeSH Terms: conditions — Respiratory System Abnormalities | interventions — Desflurane; Desmin; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desflurane (Experimental): Desflurane group: The rule of 24 will be applied, which means that the fresh gas flow (l/ min) multiplied by volume percent of desflurane must not exceed 24. Therefore, once the patients return of spontaneous ventilation, an anesthesiologist turns on oxygen 1 l/ min, nitrous oxide 1 l/ min, and desflurane 12 vol% for 1-2 minutes. When the end-tidal desflurane reaches 3-3.5% (approximately 0.5 MAC), the anesthesiologist will decrease oxygen and nitrous oxide to each 0.5 l/ min and desflurane to 6 vol% (1 MAC). Desflurane concentration will be adjusted to maintain the end-tidal desflurane around 3-6% (0.5-1 MAC).
  Interventions: Drug: Desflurane
- Sevoflurane (Active Comparator): Sevoflurane group: The oxygen and nitrous oxide each 1 l/min will be turned on with sevoflurane 4 vol% for 1-2 minutes or until the end-tidal sevoflurane reach 1-1.2% (approximately 0.5 MAC). After that, the flow of oxygen and nitrous oxide is reduced to each 0.5 l/ min and concentration dial of sevoflurane is set to 2 vol% (1 MAC). During the operation, sevoflurane concentration will be adjusted to maintain the end-tidal sevoflurane around 1-2% (0.5-1 MAC)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Desflurane — Desflurane is the volatile agent with low blood: gas partition coefficient (0.42), its uptake and elimination from the body of a patient are rapid, which results in a fast onset of anesthesia and a fast recovery from anesthesia. This property provides desflurane as an ideal agent for the ambulatory anesthesia. However, its pungent odor is concerned to irritate the upper airway and may cause significant respiratory complications.
  Other Names: Des
  Arms: Desflurane
Drug: Sevoflurane — Sevoflurane has a blood: gas partition coefficient of 0.65, which is slightly greater than desflurane. The major advantage over desflurane is the better scented. It is considered to be less airway irritation in LMA anesthesia with smooth induction and recovery.
  Other Names: Sev
  Arms: Sevoflurane

SUMMARY:
The effects of desflurane versus sevoflurane in adult patients undergoing LMA anesthesia on respiratory events during a less than 2-hour elective surgery.

DETAILED DESCRIPTION:
Laryngeal Mask Airway (LMA) anesthesia is generally performed for ambulatory surgery to avoid the use of neuromuscular blocking agents and to facilitate rapid emergence from anesthesia. Inhaled anesthetics are simply and popularly used during maintenance of anesthesia. The two most recent volatile anesthetic agents, desflurane and sevoflurane, are the two most commonly used in clinical practice for an ambulatory setting.

Desflurane is the volatile agent with low blood: gas partition coefficient (0.42). Desflurane's uptake and elimination from the body of a patient are rapid, which results in a fast onset of anesthesia and a fast recovery from anesthesia. This property provides desflurane as an ideal agent for the ambulatory anesthesia. However, its pungent odor is concerned to irritate the upper airway and may cause significant respiratory complications. Sevoflurane has a blood: gas partition coefficient of 0.65, which is slightly greater than desflurane. The major advantage over desflurane is the better scent. It is considered to be less airway irritation in LMA anesthesia with smooth induction and recovery.

The limitation of desflurane on its odor leads to a controversy if desflurane is similar to or worse than sevoflurane for LMA anesthesia. This is non-inferiority study designed to compare the occurrence of respiratory complications between desflurane and sevoflurane during LMA anesthesia.

ELIGIBILITY:
Inclusion criteria:

* Patients with American Society of Anesthesiologists physical status classification of I-III
* Elective surgery
* Surgery with expected duration of operation of less than 2 hours
* Surgery that anesthesiologist plans to use laryngeal mask airway during anesthesia

Exclusion Criteria:

* Patients with gastroesophageal reflux disease
* Patients with hiatal hernia
* Patients with history of upper respiratory tract infection within 1 month before surgery
* Heavy smoker (> 20 cigarettes per day)
* Obese patients with body mass index > 30kg/m2
* Pregnant patients
* Unable to provide a written informed consent patients
* Surgery requiring non-depolarizing muscle relaxants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of respiratory complications | From the beginning of operation until 30 minutes after the operation
  Respiratory complications are coughing, breath holding, laryngospasm, bronchospasm, and desaturation

SECONDARY OUTCOMES:
Time of eye opening | Within 30 minutes after the end of operation
  It is the time from discontinuation of anesthetic to the eye opening on verbal command.
Time to follow motor command | Within 30 minutes after the end of operation
  It is the time from discontinuation of anesthetic to hand squeezing.
Time of LMA removal | Within 30 minutes after the end of operation
  It is the time from discontinuation of anesthetic to removal of LMA.
Frequency of postoperative nausea and vomiting (PONV) | Within 2 hours after operation
  It is a number of patients with PONV in the early post-anesthetic period.
Changes of blood pressure during anesthesia | Every 15 minutes, from the beginning of operation until 30 minutes after the operation
  Non-invasive blood pressure will be recorded at the beginning of anesthesia, every 15 minutes during anesthetic maintenance, and at the time of LMA removal.
Changes of heart rate during anesthesia | Every 15 minutes, from the beginning of operation until 30 minutes after the operation
  Heart rate will be recorded at the beginning of anesthesia, every 15 minutes during anesthetic maintenance, and at the time of LMA removal.

OTHER OUTCOMES:
Time to achieve a satisfied Modified Aldrete score | Within 2 hours after operation
  It is the time that the patient is ready to be discharged from post-anesthetic care unit.
Number of Patients with high satisfaction to anesthesia | At 12-24 hour after surgery
  The satisfaction is graded using a 5-point rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Pathomporn Pin-on, M.D., Principal Investigator — Maharaj Nakorn Chiang Mai Hospital
Locations (1):
- Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
The investigators don't have a plan to share data. The investigators plan to make an individual participant data available only in site.

REFERENCES:
- [Background] de Oliveira GS Jr, Girao W, Fitzgerald PC, McCarthy RJ. The effect of sevoflurane versus desflurane on the incidence of upper respiratory morbidity in patients undergoing general anesthesia with a Laryngeal Mask Airway: a meta-analysis of randomized controlled trials. J Clin Anesth. 2013 Sep;25(6):452-8. doi: 10.1016/j.jclinane.2013.03.012. Epub 2013 Aug 17. PMID 23965188
- [Background] De Oliveira GS Jr, Fitzgerald PC, Ahmad S, Marcus RJ, McCarthy RJ. Desflurane/fentanyl compared with sevoflurane/fentanyl on awakening and quality of recovery in outpatient surgery using a laryngeal mask airway: a randomized, double-blinded controlled trial. J Clin Anesth. 2013 Dec;25(8):651-8. doi: 10.1016/j.jclinane.2013.07.006. Epub 2013 Oct 4. PMID 24095885
- [Background] Goodwin N, Strong PJ, Sudhir G, Wilkes AR, Hall JE. Effect of breathing low concentrations of volatile anaesthetic agents on incidence of adverse airway events. Anaesthesia. 2005 Oct;60(10):955-9. doi: 10.1111/j.1365-2044.2005.04279.x. PMID 16179038
- [Background] White PF, Eshima RW, Maurer A, King T, Lin BK, Heavner JE, Bogetz MS, Kaye AD. A comparison of airway responses during desflurane and sevoflurane administration via a laryngeal mask airway for maintenance of anesthesia. Anesth Analg. 2003 Mar;96(3):701-705. doi: 10.1213/01.ANE.0000048978.40522.AB. PMID 12598249
- [Background] McKay RE, Bostrom A, Balea MC, McKay WR. Airway responses during desflurane versus sevoflurane administration via a laryngeal mask airway in smokers. Anesth Analg. 2006 Nov;103(5):1147-54. doi: 10.1213/01.ane.0000237293.39466.65. PMID 17056947
- [Background] Mckay RE, Large MJC, Balea MC, Mckay WR. Airway reflexes return more rapidly after desflurane anesthesia than after sevoflurane anesthesia. Anesth Analg. 2005 Mar;100(3):697-700. doi: 10.1213/01.ANE.0000146514.65070.AE. PMID 15728054
- [Background] White PF, Tang J, Wender RH, Yumul R, Stokes OJ, Sloninsky A, Naruse R, Kariger R, Norel E, Mandel S, Webb T, Zaentz A. Desflurane versus sevoflurane for maintenance of outpatient anesthesia: the effect on early versus late recovery and perioperative coughing. Anesth Analg. 2009 Aug;109(2):387-93. doi: 10.1213/ane.0b013e3181adc21a. PMID 19608808
- [Background] Mahmoud NA, Rose DJ, Laurence AS. Desflurane or sevoflurane for gynaecological day-case anaesthesia with spontaneous respiration? Anaesthesia. 2001 Feb;56(2):171-4. doi: 10.1046/j.1365-2044.2001.01528.x. PMID 11167479